CLINICAL TRIAL: NCT03882502
Title: The Effect of Transcranial Direct Current Stimulation (tDCS) on Naming Ability in Patients With Traumatic Brain Injury Induced Aphasia
Brief Title: Electrical Stimulation in Traumatic Brain Injury (TBI) Induced Aphasia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Medicine Greifswald (Other)
Collaborators: P.A.N.-Zentrum (Other); Unfallkrankenhaus Berlin (Other); Kliniken Beelitz GmbH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: BISCUIT Trial 2019
Record Dates: First submitted 2019-03-18; First posted 2019-03-20 (Actual); Last update posted 2020-02-07 (Actual); Status verified 2020-02

CONDITIONS: Aphasia; TBI (Traumatic Brain Injury); tDCS
MeSH Terms: conditions — Aphasia; Brain Injuries, Traumatic | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- stimulation group (Experimental)
  Interventions: Other: anodal transcranial direct current stimulation (tDCS)- accompanied naming therapy or sham stimulation
- sham stimulation (Sham Comparator)
  Interventions: Other: anodal transcranial direct current stimulation (tDCS)- accompanied naming therapy or sham stimulation

INTERVENTIONS:
Other: anodal transcranial direct current stimulation (tDCS)- accompanied naming therapy or sham stimulation — anodal tDCS or sham stimulation will be combined with an intensive naming training and the number of items that could be named will be assessed immediately after the intervention.

SUMMARY:
The aim of this study is to investigate whether a tDCS-accompanied intensive naming therapy leads to a performance improvement in patients with chronic aphasia induced by a moderate TBI

ELIGIBILITY:
Inclusion Criteria:

* aphasia assessed by Aachener Aphasie Test (AAT) > 6 month after moderate TBI
* Age: 18 - 80 years
* right handedness

Exclusion Criteria:

* dementia or other neurological diseases
* History of severe alcoholism or use of drugs
* Severe psychiatric disorders such as depression, psychosis (if not in remission)
* Severe untreated medical problems such as cancer

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-07-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Naming ability assessed by | 2 weeks
  Performance in a standardised naming task (Boston Naming Task, BNT) under anodal tDCS compared to sham assessed immediately after training period

CONTACTS AND LOCATIONS:
Overall Officials: Agnes Floeel, Prof, Principal Investigator — University Medicine Greifswald
Locations (1):
- University medicine Greifswald, Greifswald, Germany